CLINICAL TRIAL: NCT06126796
Title: A Randomized Cross-Over Study to Evaluate Patient Preference and Satisfaction With Urine-based Molecular Testing Versus Cystoscopy for Surveillance of Nonmuscle Invasive Bladder Cancer (NMIBC)
Brief Title: Urine-based Molecular Testing vs Cystoscopy for Surveillance of Nonmuscle Invasive Bladder Cancer (NMIBC)
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mark D. Tyson II, M.D., M.P.H., Principal Investigator, Mayo Clinic
Other Study IDs: MDT-CxB-01; 23-008567 (Other: Mayo Clinic Institutional Review Board); NCI-2023-09278 (Registry Identifier: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Non-muscle Invasive Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — Cystoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm A: CxBladder followed by cystoscopy: Arm A will undergo testing with CxBladder 3 months after randomization followed by a cystoscopy 3 months thereafter
  Interventions: Diagnostic Test: CxBladder Monitor; Diagnostic Test: Cystoscopy
- Arm B: cystoscopy followed by CxBladder: Arm B will undergo cystoscopy 3 months after randomization followed by testing with CxBladder 3 months thereafter.
  Interventions: Diagnostic Test: CxBladder Monitor; Diagnostic Test: Cystoscopy

INTERVENTIONS:
Diagnostic Test: CxBladder Monitor — CxBladder Monitor (CxbM) is an FDA-approved genomic biomarker test specifically designed for patients undergoing surveillance for NMIBC. The non-invasive urine test quantifies 5 measured biomarker genes (MDK, HOXA13, CDC2 (CDK1), IGFBP5, CXCR2) and incorporates this information into an algorithm to detect the presence or absence of bladder cancer.
  Other Names: CxBladder; CxbM
Diagnostic Test: Cystoscopy — Cystoscopy is the most common way surveillance has been performed for NMIBC. Cystoscopy is a procedure that allows your doctor to examine the lining of your bladder and the tube that carries urine out of your body (urethra). A hollow tube (cystoscope) equipped with a lens is inserted into your urethra and slowly advanced into your bladder.

SUMMARY:
The purpose of this study is to evaluate patient-reported preference for urine based molecular testing (CxBladder Monitor) compared to cystoscopy for patients on surveillance for Nonmuscle Invasive Bladder Cancer (NMIBC). Urine based molecular testing involves noninvasive testing of a urine sample for biomarkers associated with disease recurrence. Cystoscopy is an examination of the bladder and urethra using a thin tube like instrument that is inserted into the urethra.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with a history of histologically confirmed nonmuscle invasive bladder cancer (NMIBC) who have at least 6 months of disease-free survival from last recurrence.
* Able to provide urine for testing and comply with study protocol.
* Have an email address and be willing to complete surveys online.

Exclusion Criteria:

* History of non-urothelial bladder cancer (primary squamous, adenocarcinoma, and small cell carcinoma)
* Patients with predominant (>50%) variant histology
* Patients with a history of upper tract and/or urethral cancer
* Women who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female adult patients who are undergoing cystoscopic surveillance for NMIBC after at least 9 months of recurrence-free survival.
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2023-11-16 (Actual); Primary Completion 2025-09-08 (Actual); Study Completion 2025-09-08 (Actual)

PRIMARY OUTCOMES:
Preference for CxBladder Monitor compared to cystoscopy | Up to 6 months
  Patient preference will be assessed based on the Preference Questionnaire (PQ) after completion of the study cross-over period (after both methods of testing have been experienced).

SECONDARY OUTCOMES:
Patient satisfaction | Up to 6 months
  Patient satisfaction will be assessed based on the Satisfaction Questionnaire (SQ) after completion of each test at 3 and 6 months.
Change in symptoms and function - EORTC NMIBC-24 | Up to 6 months
  The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Non-Muscle-Invasive Bladder Cancer (EORTC NMIBC-24) will be used to assess Health-related quality of life. The questionnaire consists of 24 items scored on a four-point Likert scale ranging from 1 (not at all) to 4 (very much), with the exception of the global health status items, which employ a seven-point scale ranging from 1 (very poor) to 7 (excellent). Higher scores are interpreted as more symptom burden, with exception of the sexual function and sexual enjoyment sections, where higher scores represent better functioning.
Fear of Cancer Recurrence Inventory- Short Form (FCRI-SF) | Up to 6 months
  Health-related quality of life will be assessed based on the Fear of Cancer Recurrence Inventory- Short Form (FCRI-SF) at baseline, 3 months (within 1 week of test), and 6 months (within 1 week of test). The nine-item FCRI evaluates the presence and severity of intrusive thoughts associated with FCR. Each item is rated on a Likert scale ranging from 0 ("not at all" or "never") to 4 ("a great deal' or "all the time"). A higher score indicates higher levels of FCR.
Financial costs | Up to 6 months
  Assessed by patient responses to questions about missed work and time missed from usual activities.
Error rate identifying recurrent nonmuscle invasive bladder cancer (NMIBC) | Up to 6 months
  Error rate for CxBladder is defined as the proportion of patients who have a negative CxBladder at 3 months but have a recurrence identified on cystoscopy at 6 months for patients in arm A. The error rate for cystoscopy is defined as the proportion of patients who have a negative cystoscopy at 3 months but have a positive CxBladder at 6 months that is subsequently confirmed by cystoscopy for patients in arm B.

CONTACTS AND LOCATIONS:
Overall Officials: Mark D. Tyson, M.D., M.P.H., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials